CLINICAL TRIAL: NCT04118582
Title: Resting Metabolic Rate: is a Predictor Weight Regain?
Brief Title: Resting Metabolic Rate is a Predictor of Weight Regain?
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Roberto de Cleva, Principal investigator, University of Sao Paulo General Hospital
Other Study IDs: 00984812.5.0000.0068
Record Dates: First submitted 2019-04-30; First posted 2019-10-08 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Severe Obesity
Keywords: severe obesity; resting metabolic rate; indirect calorimetry; body composition; electrical bioimpedance analisys
MeSH Terms: conditions — Obesity, Morbid | interventions — Body Composition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective analisys: Bioimpedance The BC measurements as FM (% and kg), FFM (% and kg), will be obtained by the indirect noninvasive method of electrical bioimpedance (BIA) 230, 2.0, (Biospace Seoul, Korea). Those evaluated will be standing and positioned on the platform electrodes, barefoot and with their arms extended with their hands on the two supports (electrodes).
  Evaluation of RMR For the evaluation of the RMR, the values of VO2 and VCO2 will be collected by the indirect calorimetry (IC) method using the Ultima CPX metabolic analyzer (MedGraphics, USA), calibrated with each test.
  Interventions: Other: Body composition and resting metabolic rate analisys

INTERVENTIONS:
Other: Body composition and resting metabolic rate analisys

SUMMARY:
he increasing prevalence of obesity in developed countries has also reached Brazil in the last two decades. Conventional treatments are not efficient to sustained weight loss and in some cases, weight reduction in individuals refractory to these methods. Bariatric surgery has been considered as the most efficient long-term treatment. However, numerous studies have reported weight regain in approximately 20% of patients, from the second year of surgery. The objective of this study is to analyze the changes in resting metabolic rate and body composition before, 6 and 36 months after weight loss and its relation to late weight regain. 48 adults of both sexes, above 18 years, will undergo bypass performed the ambulatory of the Bariatric and Metabolic Surgery Unit of the Department of Gastroenterology of HCFMUSP. Patients over 60 years, undergoing revision surgery and other surgical techniques will be excluded. The body weight (kg) will be measured by In Body 230. BMI (kg/m2) shall be determined by dividing body weight (kg) by height (m) squared. Excess weight (kg): difference in preoperative weight versus ideal weight considered for weight for BMI 25kg/m2. Weight loss (kg): pre-surgery weight difference in relation to the lowest weight reached after 18 months. Percentage of excess of weight loss is difference of weight loss in relation to overweight, used as an indicator of success of surgery. Fat mass (%, kg) and fat-free mass (%, kg) will be obtained by electrical bioimpedance 230, 2.0. For resting metabolic rate, the values of VO2 and VCO2 will be collected by indirect calorimetry using Ultima CPX metabolic analyzer. The daily energy expenditure (kcal/day) will be calculated by the Weir equation.

keywords: obesity, resting metabolic rate, body composition analysis, bariatric surgery.

DETAILED DESCRIPTION:
INTRODUTION The increasing prevalence of obesity in developed countries has also reached Brazil in the last two decades and is now among the ten countries with the largest number of obese people in the world1.

According to the Vigilance Survey of Risk Factors and Protection for Chronic Diseases by Telephone Inquiry (Vigitel, 2014), overweight in Brazil affects 49.1% of women and obesity affects 18.2% of male population2.

The most recent data on the spread of the disease in the world present alarming numbers. It is estimated that 1.9 billion adults around the world are overweight and more than 600 million are considered obese3.

Characterized by excess of body fat, obesity is a chronic disease of multifactorial origin that is difficult to handle when it reaches body mass index (BMI) above 40 kg/m2. In these cases, conventional treatments such as restriction food intake, medication and monitored physical exercise are not efficient to sustained weight loss and in some cases, weight reduction in individuals refractory to these methods4.

For those individuals who do not respond to these treatments for more than two years and BMI ≥35 kg/m2 with comorbidities such as sleep apnea, Type 2 Diabetes Mellitus, hypertension, dyslipidemias, depression, asthma, infertility among others, surgery has been considered as the most efficient long-term treatment. Surgical treatment results in loss of between 20 and 40% of the initial weight or between 60 and 80% of the excess weight, as well as higher rates of remission of Type 2 Diabetes and Metabolic Syndrome, improvement in the quality of life and reduction in use hypoglycemic, antihypertensive and hypolipidemic drugs5-7.

However, numerous studies have reported weight regain in approximately 20% of these patients, from the second year of surgery. The review by Shah et al. demonstrates long-term weight loss and the risk of recurrence of obesity-related comorbidities8. Similar results were observed in the study by Pajecki et al. when evaluated between 5 and 9 years after surgery9.

Weight recovery has been justified by a variety of causes, such as the surgical method used, especially those that are strictly restrictive, the technical failure of the operation and the eating behavior, influenced or not by mental health factors such as anxiety, depression, binge eating. More recently, it has been discussed possible failures in entero-hormonal stimulation that could influence the reduction of satiety as demonstrated by Santo et al10,11.

Another hypothesis for weight regain would be the reduction of metabolic rate due to massive weight loss. Das et al. observed a 25% drop in resting energy expenditure after weight loss and stabilization due to loss of free fat mass and fat mass suggesting that there was a metabolic adaptation and an increase in energy efficiency when evaluated after 14 and 24 months12.

The association of weight loss and marked fall in the resting metabolic rate (RMR) probably occurs due to thermogenic adaptation, since the loss of 10% or more of body weight (BW) can reduce the energy expenditure of 24h by approximately 20-25%. Thus, the energy needs fall by 300-400 calories/day for weight maintenance is 10-15% lower when compared to a non-obese individual, based only on FFM and FM reduction13,14.

Bariatric surgery is associated with a decrease in total energy expenditure due to a reduction in the resting metabolic rate, which may be justified by the alteration of the body composition (BC) of both FFM and FM15.

For Abdeen and Roux, patients regaining weight after 2 years had low resting energy expenditure after RYGB and the decrease in metabolic rate can be attenuated when the relative lean mass preservation occurs16. However, in this same review, in the study by Carrasco et al. it could be observed that the drop in energy expenditure/FFM% was positively related to the initial energy expenditure and to the change in the percentage of FM, indicating that the metabolic adaptation was not associated with loss of FFM but with high RMR before surgery17.

Olbers et al. observed the reduction in the RMR of 50 individuals submitted to gastric bypass and vertical gastroplasty after one year and did not find a statistical difference when compared between the different surgical techniques18.

The study conducted by Faria et al. evaluated the RMR of 36 patients after two years of surgery, separating them into two groups. The group of individuals who had recovered from 2 kg of the total weight presented an average difference of 260 kcal/day lower than the group that maintained the weight. When RMR was calculated from predictive equations it was observed that they are overestimated in this weight regimen19.

Although the impact of diet-induced weight loss on energy expenditure has been widely studied, the impact of bariatric surgery on total energy expenditure, resting energy expenditure, and diet-induced thermogenesis has not yet been fully elucidated. A compelling hypothesis would be the modification of the BCn20.

The Centers for Disease Control and Prevention (CDC) recommends the Body Mass Index (BMI), where weight (kg)/height (m)2, as a reference for the diagnosis of obesity, using different classifications to determine the degrees of severity of disease. However, although its use is widely diffused due to its simple applicability, either in ease of measurement or in the minimum cost, it is considered an imprecise measure since it does not consider the great variation of fat distribution and the body components such as FM, FFM, muscle mass, bone mass and water21,22.

The precise evaluation of the BC through the determination of its components allows establishing prognostic of the occurrence of diseases associated with the high amount of corporal fat. It would also be possible to establish interventions with adequate evaluation of body compartment alterations, especially after surgical treatment of obesity, where weight loss occurs intensely and leads to a change in BC23-26.

In the study by Flanbaum et al. the group of patients stratified as hypometabolic presented a significant increase in the metabolic rate in the first six weeks post-bypass, while there was no change in the normometabolic group. This pattern changed significantly in reevaluation after 2 years, when the normometabolic group had a reduction in the resting metabolic rate, although it remained within the normality norm, indicating a compensatory metabolic response to the food restriction designed to "protect" body weight27.

The maintenance of basic body activities is represented by RMR or resting energy expenditure28. RMR can be defined as the energy required by the body at rest or the amount of energy spent by the individual while awake after an absorptive period in a thermally neutral environment and without having exercised in the last 24 hours29.

RMR and basal metabolic rate (BMR) are similar and differ only in gauging, since BMR is measured in the morning, after a fasting night, without any exercise in the last 24 hours, free of emotional stress, familiarized with the appliance and completely rested30. In general, RMR may be a better indicator of daily energy requirements than RMR31.

RMR is slightly larger than BMR, since it adds to the latter the additional energy expenditure required for muscle contraction. However, it differs from the former by less than 10%, allowing both to be used. Representing the main component of daily energy expenditure, RMR corresponds to 60% to 75% of total expenditure and in active individuals can reach 50%32-34. while in sedentary individuals, up to 75%. Dietary energy expenditure, when macronutrient absorption occurs, lasts around 12 hours after the last meal, corresponds to approximately 10%, and energy expenditure with physical activity (acute or chronic) is not included. between 15% and 30% (Figure 1)32-34.

The determination of RMR depends to a large extent on the amount of muscle mass and the activity of other metabolically active tissues such as heart, brain, kidneys and liver35.

Figure 1. The thermodynamic perspective of energy expenditure

Bradford B. (2000)36 In a meta-analysis conducted by McMurray et al. comparative studies on the influence of sex, age and nutritional status on RMR have recently been identified. African Americans had approximately 10% to 20% lower RMR than whites and lower FM than in Caucasians or Hispanics. Among women, rates are lower than in men and in the elderly lower than in young adults. Differences between gender and age groups could be related to the composition of FFM, a metabolically more active tissue, mainly muscle mass37. In addition, the literature on RMR is clear about the location of FM in the body, important for its understanding38.

Studies have shown that FM can influence RMR as well as muscle mass, especially when it is predominantly located in the abdominal region, which indicates that it also has a metabolic function when compared to total fat. The study by Luhrmann evaluated the relationship between abdominal and peripheral fat with MRT and demonstrated that abdominal fat influenced in women39.

Visceral fat is metabolically more active than the others because it is associated with the release of free fatty acids in the portal circulation which can lead to peripheral hyperinsulinemia and, therefore, less sensitivity to its anti-lipolytic effect. Visceral fat plays a predominant role in the development of metabolic complications, in addition to justifying the correlation between central fat and RMR40-42.

JUSTIFICATION The relevance of this study is to identify/analyze the changes in RMR and BC after bariatric surgery and its relation to weight regain.

OBJECTIVE To analize RMR and body composition (FM, FFM) before and after weight loss (6 and 36 months) induced by bariatric surgery with weight regain.

METHODS Ethic This study was elaborated and will be performed at the Clinical Hospital of the Medical School of the University of São Paulo (HCFMUSP). The patients involved will receive the Informed Consent Form (ICF) for their agreement to participate in the study.

Study Prospective study keywords: obesity, resting metabolic rate, body composition analysis, bariatric surgery.

Casuistic The sample, calculated through Test t (Annex 1), consists of 49 adults selected at the ambulatory of the Bariatric and Metabolic Surgery Unit of the Department of Gastroenterology of HCFMUSP in the periods: preoperative, 6 and 36 months after surgery.

Inclusion criteria Patients of both sexes, above 16 years of age, will undergo bypass techniques and vertical gastroplasty performed at the institution.

Exclusion Criteria Adult patients over 60 years old, undergoing revision surgery and other surgical techniques will be excluded.

Anthropometric Assessment Anthropometric variables will be obtained on the same day as the evaluation of BC by trained evaluators.

The PC body weight (kg) will be measured by In Body 230, 2.0, (Biospace Seoul, Korea). The patient should be in the orthostatic position, facing the display, in the center of the scale, barefoot, in light clothes.

The height measurement (m) will be performed in a stadiometer coupled to the scale W 300, Class III, with a maximum capacity of 2m. The patient will be kept with his back to the meter, with the feet united, in an erect position, looking at horizon and arms extended to the side of the body. The reading will be made in the nearest centimeter when the horizontal rod of the vertical bar of the stature scale rests against the individual's head.

BMI (kg/m2) shall be determined by dividing body weight (kg) by height (m) squared.

Excess weight (EW, kg): difference in preoperative weight versus ideal weight. The ideal weight (IW, kg) considered for the calculation of weight regain will be weight for BMI 25kg/m2.

Weight loss (WL, kg): pre-surgery weight difference in relation to the lowest weight reached after 18 or 24 months, obtained through the medical record.

Percentage of excess of weight loss (% EWL): percentage difference of weight loss in relation to overweight, used as an indicator of success of surgery43.

Evaluation of BC and RMR The evaluations will be held between 8:00 am and 10:00 am in the Laboratory of Exercise and Movement Studies at the Institute of Orthopedics and Traumatology of FMUSP.

Bioimpedance The BC measurements as FM (% and kg), FFM (% and kg), will be obtained by the indirect noninvasive method of electrical bioimpedance (BIA) 230, 2.0, (Biospace Seoul, Korea). Those evaluated will be standing and positioned on the platform electrodes, barefoot and with their arms extended with their hands on the two supports (electrodes).

Evaluation of RMR For the evaluation of the RMR, the values of VO2 and VCO2 will be collected by the indirect calorimetry (IC) method using the Ultima CPX metabolic analyzer (MedGraphics, USA), calibrated with each test. The daily energy expenditure (kcal/day) will be calculated by the Weir equation44.

Equation Weir = [(3,9 * O2) + (1,1 * CO2) * 1440], where: O2 is the mean value consumed (L/min) and CO2 is the expired mean value (L/min) 20 minutes computed for analysis.

For the day before the test day patients will be instructed to avoid drinking coffee, alcohol or stimulants. For the test, they will be advised to wear light and comfortable clothing, to fast from 4 h to 6 h and to make minimal physical effort on the way to the laboratory on the test day. During the test, the patient should remain supine, avoid moving or sleeping.

The test will be performed under laboratory conditions for 40 min, and the spirometric values will be collected from respiration to respiration. To begin the computation of the data, with the individual already connected to the metabolic analyzer, data from the initial 20 minutes for the stability of the physiological variables at rest will be neglected.

RMRs will be calculated from the BIA and the Milflin's equation45. Evaluation of parameters laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes,
* Above 18 to 60 years

Exclusion Criteria:

* Adult patients over 60 years old,
* patients undergoing revision surgery and other surgical techniques will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample consists of 48 adults, both sexes, BMI > 40 kg/m² < 60 kg/m², selected at the ambulatory of the Bariatric and Metabolic Surgery Unit of the Department of Gastroenterology at the Clinical Hospital of the Medical School of the University of Sao Paulo (HCFMUSP).
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in resting metabolic rate | Before, 6 months and 36 months after bariatric surgery
  This will be evaluated by indirect calorimetry before and after bariatric surgery: kcal per day and per kilogram fat free mass.
Late weight regain | 18 months of bariatric surgery
  This will be evaluated considering the lowest weight (in kilos) reached after 18 months of bariatric surgery
Changes in body composition | Before, 6 months and 36 months after bariatric surgery
  This will be evaluated fat mass (kg, %) and fat-free mass (kg,%) by electrical bioimpedance before and after 6 and 36 months of bariatric surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto de Cleva, MD PhD, Study Chair — Clinical Hospital of University of Sao Paulo Medical School; Lilian Cardia, MsC, Principal Investigator — University of Sao Paulo Medical School
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo, Brazil

REFERENCES:
- [Background] Santo MA, Riccioppo D, Pajecki D, Kawamoto F, de Cleva R, Antonangelo L, Marcal L, Cecconello I. Weight Regain After Gastric Bypass: Influence of Gut Hormones. Obes Surg. 2016 May;26(5):919-25. doi: 10.1007/s11695-015-1908-z. PMID 26450709
- [Background] Browning MG, Franco RL, Cyrus JC, Celi F, Evans RK. Changes in Resting Energy Expenditure in Relation to Body Weight and Composition Following Gastric Restriction: A Systematic Review. Obes Surg. 2016 Jul;26(7):1607-15. doi: 10.1007/s11695-016-2184-2. PMID 27103027
- [Background] Faria SL, Faria OP, Cardeal Mde A, de Gouvea HR, Buffington C. Diet-induced thermogenesis and respiratory quotient after Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2012 Nov-Dec;8(6):797-802. doi: 10.1016/j.soard.2012.06.008. Epub 2012 Jul 23. PMID 22884301
- [Background] Flancbaum L, Verducci JS, Choban PS. Changes in measured resting energy expenditure after Roux-en-Y gastric bypass for clinically severe obesity are not related to bypass limb-length. Obes Surg. 1998 Aug;8(4):437-43. doi: 10.1381/096089298765554331. PMID 9731680